CLINICAL TRIAL: NCT02974777
Title: Individualizing Dual Antiplatelet Therapy After Percutaneous Coronary Intervention - The IDEAL-PCI Extended Registry
Brief Title: The IDEAL-PCI Extended Registry
Acronym: IDEAL-PCI ext
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: not started due to regulatory reasons
Sponsor: Kaiser Franz Josef Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Guenter Christ, Prof, Kaiser Franz Josef Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDEAL-PCI v.2
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Coronary Arterioscleroses; Platelet Dysfunction Due to Drugs
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- Bleeding prevention group (Active Comparator): Patients with reduction of standard dose DAPT due to low platelet reactivity to asprin and/or P2Y12 inhibitor
  Interventions: Drug: DAPT reduction; Drug: DAPT on-target
- Ischemia prevention group (Active Comparator): Patients with intensification of standard dose DAPT due to high platelet reactivity to asprin and/or P2Y12 inhibitor
  Interventions: Drug: DAPT on-target; Drug: DAPT intensification

INTERVENTIONS:
Drug: DAPT reduction — Reduction of standard dose DAPT due to low platelet reactivity
  Arms: Bleeding prevention group
Drug: DAPT on-target — Standard DAPT within the therapeutic window of platelet reactivity
Drug: DAPT intensification — Intensification of standard dose DAPT due to high platelet reactivity
  Arms: Ischemia prevention group

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a routine individualized antiplatelet therapy after coronary stent implantation by evaluating "on-treatment" platelet reactivity with Multiple Electrode Aggregometry (MEA, Multiplate® Analyzer).

IDEAL-PCI Extended is the continuation of the IDEAL-PCI registry with additional focus on bleeding events and net clinical benefit

DETAILED DESCRIPTION:
Determination of platelet reactivity in patients with percutaneous coronary Intervention as described in the IDEAL-PCI registry.

In the IDEAL-PCI Extended Registry an additional deescalation arm with reduction of the standard dual antiplatelet therapy (DAPT) dosis in case of low platelet reactivity to P2Y12 Inhibition or Aspirin with or without bleeding is implemented.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive PCI patients

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
stent thrombosis | 1 year
  stent thrombosis by any Academic Research Consortium (ARC) definition
bleeding | 1 year
  bleeding type 1-3 and 5 by Bleeding Academic Research Consortium (BARC) definition

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular Events (MACCE) | 1 year
  death, cardiovascular death, myocardial infarction, stroke, ischemia driven revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Christ, MD, Principal Investigator — Kaiser Franz Josef Hospital
Locations (1):
- Kaiser Franz Josef Hospital, Vienna, Austria

REFERENCES:
- See also: IDEAL-PCI Registry — http://clinicaltrials.gov/ct2/show/NCT01515345